CLINICAL TRIAL: NCT00921167
Title: A Phase II Study to Evaluate the Efficacy of Bevacizumab Plus Irinotecan in Recurrent Anaplastic Astrocytoma or Recurrent Glioblastoma Multiforme
Brief Title: A Study to Evaluate the Efficacy of Bevacizumab Plus Irinotecan in Recurrent Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Research Center for Solid Tumor, Korea (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L-0006
Record Dates: First submitted 2009-06-13; First posted 2009-06-16 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Glioblastoma; Astrocytoma
Keywords: Glioblastoma; Astrocytoma; Chemotherapy
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab/Irinotecan (Experimental)
  Interventions: Drug: Bevacizumab/Irinotecan

INTERVENTIONS:
Drug: Bevacizumab/Irinotecan — Bevacizumab 10mg/kg D1 Irinotecan 125mg/m2 D1 (without enzyme-inducing antiepileptic drugs [EIAEDs] or 340mg/m2 for patients on EIAEDs) every 2 weeks

SUMMARY:
To assess the efficacy and safety of bevacizumab plus irinotecan for the patients with recurrent anaplastic astrocytoma or with recurrent glioblastoma multiforme

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed recurrent anaplastic astrocytoma or recurrent glioblastoma multiforme
* At least 18 years of age
* Performance status of 0 and 1 on the Eastern Cooperative Oncology Group (ECOG) criteria
* One or more measurable disease
* Adequate hematologic (neutrophil count >= 1500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit (UNL)x2.5, bilirubin level =< UNLx1.5, alkaline phosphatase =< UNLx2.5), and renal (creatinine clearance >= 30mL/min)
* Expected life time more than at least 2 months
* A patients who signed the informed consent prior to the participation in the study

Exclusion Criteria:

* A pregnant or lactating patient
* A patient of childbearing potential without being tested for pregnancy at baseline or with a positive test. (A premenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
* A man or woman of childbearing potential without the willingness to use a contraceptive measures during the study
* A patient with history of another malignant disease within past 3 years, except curatively treated basal cell carcinoma of the skin, cervical carcinoma in situ, and early gastric cancer
* Medically uncontrolled serious heart, lung, neurological, psychological, or metabolic disease
* Uncontrolled serious infection
* Enrollment in other study within 30 days
* Hemorrhage on baseline radiologic examination
* A patient who refused to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months, 1 year

SECONDARY OUTCOMES:
Objective response rate | 6 weeks, 12 weeks
Overall survival | 6 months, 1 year
Disease-control rate | 6 weeks, 12 weeks
Adverse event | 3 weeks, 6 weeks, 9 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea